CLINICAL TRIAL: NCT06998628
Title: Clinical Study Evaluating the Effect of Pentoxifylline as Anti Inflammatory in Patients With Rheumatoid Arthritis
Brief Title: Pentoxifylline as Anti-Inflammatory in Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Prof. Sahar Kamal Hegazy, Professor of Clinical Pharmacy, Faculty of Pharmacy - Tanta University (Unknown); Dr. Mustafa Adel Mustafa Elmenawy Lecturer of Rheumatology and Rehabilitation, Faculty of Medicine - El-Azhar University - Damietta (Unknown)
Responsible Party: Principal Investigator, Shrouk Ali Mohamed Elsies, Demonstrator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 78956
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): will receive the traditional therapy of RA for three months.
  Interventions: Drug: Methotrexate
- Pentoxifylline group (Active Comparator): will receive 400 mg pentoxifylline two times daily plus the traditional therapy of RA for three months.
  Interventions: Drug: Methotrexate; Drug: Pentoxifylline

INTERVENTIONS:
Drug: Methotrexate — Methotrexate (MTX) is a chemotherapy agent and immune-system suppressant. It is used to treat cancer, autoimmune diseases, and ectopic pregnancies. Types of cancers it is used for including breast cancer, leukemia, lung cancer, lymphoma, gestational trophoblastic disease, and osteosarcoma. Methotrexate is also used to treat rheumatoid arthritis and other inflammatory conditions.
Drug: Pentoxifylline — Pentoxifylline (also known as oxpentifylline) is a methylxanthine derivative with strong hemorrheologic effects. In the United States, it is primarily used to treat intermittent claudication. Studies in both humans and animals have demonstrated that pentoxifylline therapy induces various physiological changes at the cellular level
  Arms: Pentoxifylline group

SUMMARY:
Rheumatoid arthritis (RA) is a long-term inflammatory condition that leads to gradual damage of joints lined by synovial membranes, along with various potential effects outside of the joints. While RA can affect any joint, it typically involves the metacarpophalangeal, proximal interphalangeal, and metatarsophalangeal joints, as well as the wrists and knees. Symptoms related to the joints and surrounding tissues include swelling, tenderness upon touch, morning stiffness, and significant difficulty moving the affected joints

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis (not in remission) according to American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) [9] i.e., 28 joints disease activity score (DAS 28) >2.6.
* Patients receiving the conventional DMARDs.
* Both sexes.
* Age range between 18and 70 years old

Exclusion Criteria:

* Patients with retinal or cerebral hemorrhage.
* Patients with renal and hepatic dysfunction.
* Patients with hypersensitivity to study medications.
* Pregnant and lactating females.
* Patients receiving biological or synthetic DMARDs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
change in Disease Activity Score (DAS28) | 3 months
  Calculation of 28-joint count Disease
  Activity Score (DAS28) using C- reactive protein level (CRP) according to the following formula:
  DAS28-CRP = [0.56*√ (tender joint count) + 0.28*√ (swollen joint count) + 0.36*ln (CRP+1)]
  *1.10 + 1.15] will be done where sever disease activity ≥ 5.1, moderate disease activity from 3.2 to 5.1, mild disease activity from 2.6 to 3.2, and remission <2.6.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Al-Azhar University, Damietta, Damietta Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No